CLINICAL TRIAL: NCT05256056
Title: Comparison of the Volume Dependent Effect of Pericapsular Nerve Block in Patients Operated for Femur Fracture: A Randomized Prospective Study
Brief Title: Volume Dependent Effect of Pericapsular Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gamze Dilara Demir, specialist medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/516
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Post Operative Pain; Femur Fracture
Keywords: pericapsular nerve group block; femur fracture; postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative; Femoral Fractures | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Group A patients will be injected with 20 cc of 0.25% Bupivacaine, and Group B patients will be injected with 30 cc of 0.25% Bupivacaine
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be randomized using the closed envelope method. While the practitioner knows the interventions to be made, the data collector will collect the data without learning the patient's group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): patients will be injected with 20 cc of 0.25% Bupivacaine
  Interventions: Drug: Bupivacain
- Group B (Experimental): patients will be injected with 30 cc of 0.25% Bupivacaine.
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — efficacy of bupivacaine in different volumes

SUMMARY:
In PENG block technique, the local anesthetic agent is injected between the psoas tendon and the pubic ramus to block the sensory branches of the nerves which innervates the hip capsule for providing analgesia without causing muscle weakness. Since the PENG block is a facial plane block, it causes a volume dependent distribution. There are a few case reposts and cadaveric studies on volume dependent effect of analgesia and motor weakness of PENG block.

In our study, we aimed to evaluate the clinical effects of the volume-dependent efficacy of PENG block.

DETAILED DESCRIPTION:
Femur fracture is the one of the most common case groups and it is seen mostly in the elderly patient population with comorbidities. For these patients, perioperative, postoperative analgesia and early mobilization are important to reduce cardiopulmonary complications and morbidity. Femoral fracture operations are mostly performed under spinal anesthesia especially under unilateral spinal anesthesia to sustain more stable hemodynamics. The lateral decubitus position, which is used for unilateral spinal anesthesia, is a painful position for these patients. Intravenous opioids are used for this procedure, however they have possible side-effects, such as sedation, inhibition of respiratory, lower blood pressure. Because of these reasons, pericapsular nerve block (PENG) has been applied recently to avoid complications. By using PENG block , positioning for spinal anesthesia is easier for patients and anesthesiologists, and postoperative analgesia can be provided.

By PENG block, the local anesthetic agent is injected between the psoas tendon and the pubic ramus to block the sensory branches of the nerves innervating the hip capsule, thus providing analgesia in patients, but muscle weakness is not expected. Becacuse PENG block is a facial plane block, it shows a volume dependent distribution. There are a few case reposts and cadaveric studies, which are showing volume depend effect of analgesia and motor weakness of PENG block.

In our study, we aimed to evaluate the clinical effects of the volume-dependent efficacy of PENG block.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergoing hip arthroplasty surgery
* Patients over the age of 18
* ASA I-II-III patients
* Patients who will be operated under spinal anesthesia

Exclusion Criteria:

* ASA IV patients, Pregnant women
* Patients who are not suitable for spinal anesthesia
* Patients diagnosed with Alzheimer's and dementia who cannot cooperate
* Patients who are not suitable for peripheral nerve block (patients with infection in the injection area, with local anesthetic allergy, with coagulopathy)
* Patients who do not want to participate in the study
* Patients under the age of 18
* Patients switched to general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
visual analouge scale | up to 24 hours,
  the VAS 0 means no pain, 10 means the worst pain possible
pin-prick test | up to 20 minutes
  the ability to determine the difference between sharp and dull.

SECONDARY OUTCOMES:
cold sensation test | up to 20 minutes
  feel the cold: 0, not feel : 1
presence of quadriceps motor block | up to 24 hours
  Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).

CONTACTS AND LOCATIONS:
Overall Officials: leyla kılınç, Study Chair — şişli etfal eğitim araştırma hastanesi
Locations (1):
- Sisli Etfal Research and Training Hospital, Seyrantepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pascarella G, Costa F, Del Buono R, Pulitano R, Strumia A, Piliego C, De Quattro E, Cataldo R, Agro FE, Carassiti M; collaborators. Impact of the pericapsular nerve group (PENG) block on postoperative analgesia and functional recovery following total hip arthroplasty: a randomised, observer-masked, controlled trial. Anaesthesia. 2021 Nov;76(11):1492-1498. doi: 10.1111/anae.15536. Epub 2021 Jul 1. PMID 34196965
- [Background] Sandri M, Blasi A, De Blasi RA. PENG block and LIA as a possible anesthesia technique for total hip arthroplasty. J Anesth. 2020 Jun;34(3):472-475. doi: 10.1007/s00540-020-02768-w. Epub 2020 Mar 30. PMID 32232662